CLINICAL TRIAL: NCT00340743
Title: Inhibition of Fried Meat-Induced DNA Damage: A Dietary Intervention Study
Brief Title: Diet and Genetic Damage
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904169; 04-E-N169
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07-16

CONDITIONS: Diet
Keywords: Heterocyclic Aminos; Cruciferous Vegetables; Yogurt; Chlorophyllin; Comet Assay; Diet; Healthy Volunteer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
This study will examine the risks and protective effects of dietary factors on temporary genetic damage to cells lining the gastrointestinal tract and to blood cells. Some foods, including very well done meat, may increase genetic damage in cells, while others, such as yogurt and vegetables, may reduce genetic damage. This study may provide new information on the influence of diet on increasing or decreasing the risk of developing cancer, particularly colorectal cancer. The study is conducted at the General Clinical Research Center (GCRC) of the University of North Carolina.

Nonsmoking, English-speaking, healthy adults between 18 and 45 years of age may be eligible for this 4-week study. Participants undergo the following tests and procedures:

* Interview: Participants complete questionnaires including information on their diets, habits, past and present health, and family histories.
* Diet: Participants adhere strictly to the diet provided by the dietician at the GCRC for all 4 weeks of the study. All meals are provided by the GCRC. All meals contain well-done meat and some contain yogurt, cruciferous vegetables, including broccoli and cabbage, and chlorophyllin tablets. Chlorophyllin is a compound in some foods that protects against genetic damage.
* Urine sampling: Participants collect a urine sample each morning except Saturday and Sunday.
* Stool sampling: Participants collect two stool samples during the study, one during the second week and another during the fourth week.
* Blood draw: About 2-1/2 tablespoons of blood are drawn once a week for research purposes. The blood is tested for the effects of eating foods in the different diets used in the study.
* Rectal biopsies: Four pinch biopsies, each about the size of a grain of rice, are taken from the rectum once a week for research purposes. For this procedure, forceps are inserted shallowly into the rectum to collect the tissue. The effects of the different diets on the colon cells are measured.

DETAILED DESCRIPTION:
Colorectal cancer is one of the most common forms of cancer worldwide and is the second leading cause of cancer death in the United States. Given the frequency of occurrence and the poor prognosis for many afflicted individuals, prevention of this disease has been a major public health priority for the past few decades. However evidence from epidemiological studies has yet to explain the tremendous excess risk in developed countries, a trend that has been tentatively attributed to lifestyle and dietary factors. In the past few years, the consumption of red meat in particular, and other meat products, has attracted considerable attention in epidemiological, clinical, and experimental studies, with an increasing focus on a certain class of compounds found in cooked meat, heterocyclic amines. Heterocyclic amines are substances formed through pyrolysis of amino acids and creatine when meats are cooked at high temperature, particularly by pan-frying. Heterocyclic amine levels increase with cooking temperature, with the type and shape of the cooked piece of meat, with the degree of browning on the surface, and with the cooking method. In several epidemiological studies, including studies from Harvard, the International Agency for Research on Cancer (IARC), and the National Cancer Institute (NCI), individuals with long-term exposure to heterocyclic amines in their diet had an increased risk of colorectal cancers and colorectal adenomas, respectively. However, not all studies of heterocyclic amines in humans have shown a positive association with colorectal cancer risk, and clear consensus regarding this association is lacking. Based on the implications from these epidemiological studies, researchers at NCI have recently conducted a series of controlled feeding studies aimed at relating short-term exposure to heterocyclic amines through fried meat consumption to transient changes in urine mutagenicity levels. These studies provide evidence that meat fried at high temperatures results in significant short-term increases in exposure to mutagens. However, whereas urine mutagenicity appears to be a good short-term measure of exposure to heterocyclic amines in the diet, it is unclear as to whether these compounds induce genetic damage in colonic epithelial cells in humans. Against this background, we propose conducting a feeding study that includes the examination of colon tissue for evidence of transient DNA damage detected in the single cell gel electrophoresis (comet) assay following experimental intake of fried meat. This study will provide more direct evidence than previous studies as to whether genetic damage in colon epithelium and lymphocytes is related to dietary intake of heterocyclic amines. The use of the comet assay to detect the effects of diet on transient DNA damage is novel in this type of controlled feeding study, particularly with respect to monitoring effects of diet on colon epithelial cells. We will also monitor effects of fried meat ingestion on DNA damage in lymphocytes and detect changes in urinary mutagenicity related to these dietary regimens.

ELIGIBILITY:
* INCLUSION CRITERIA:

Nonsmoking, English speaking, healthy adults, ages 18-45 will be enrolled.

EXCLUSION CRITERIA:

Pregnant women will be excluded, as the dietary regimen in this study is not optimal for pregnant women.

Individuals will also be excluded if they consume more than two alcoholic drinks per day, have a history of illicit drug use, have a history of goiter, diabetes, colitis, or a diagnosed current thyroid condition, are excessively obese (BMI greater than 30), are vegetarians, or are currently taking anti-coagulant medication.

Individuals on prescription medications or antibiotics will be excluded.

Consumption of tea, or use of aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), or vitamin or herbal supplements by participants will also be prohibited during the study.

Alcohol consumption will be prohibited during the study.

Children will not be enrolled in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2004-04-21; Study Completion 2019-07-16

PRIMARY OUTCOMES:
to determine if eating certain foods and other dietary constituents will ameliorate the short-term damaging effects associated with fried meat consumption. | Continuously

CONTACTS AND LOCATIONS:
Overall Officials: Jack Taylor, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Butler LM, Sinha R, Millikan RC, Martin CF, Newman B, Gammon MD, Ammerman AS, Sandler RS. Heterocyclic amines, meat intake, and association with colon cancer in a population-based study. Am J Epidemiol. 2003 Mar 1;157(5):434-45. doi: 10.1093/aje/kwf221. PMID 12615608
- [Background] Baker R, Arlauskas A, Bonin A, Angus D. Detection of mutagenic activity in human urine following fried pork or bacon meals. Cancer Lett. 1982 May-Jun;16(1):81-9. doi: 10.1016/0304-3835(82)90094-5. PMID 6811131
- [Background] DeMarini DM, Hastings SB, Brooks LR, Eischen BT, Bell DA, Watson MA, Felton JS, Sandler R, Kohlmeier L. Pilot study of free and conjugated urinary mutagenicity during consumption of pan-fried meats: possible modulation by cruciferous vegetables, glutathione S-transferase-M1, and N-acetyltransferase-2. Mutat Res. 1997 Nov 19;381(1):83-96. doi: 10.1016/s0027-5107(97)00152-8. PMID 9403034
- [Derived] Shaughnessy DT, Gangarosa LM, Schliebe B, Umbach DM, Xu Z, MacIntosh B, Knize MG, Matthews PP, Swank AE, Sandler RS, DeMarini DM, Taylor JA. Inhibition of fried meat-induced colorectal DNA damage and altered systemic genotoxicity in humans by crucifera, chlorophyllin, and yogurt. PLoS One. 2011 Apr 25;6(4):e18707. doi: 10.1371/journal.pone.0018707. PMID 21541030